CLINICAL TRIAL: NCT06748079
Title: Phase I Clinical Study on the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Characteristics of Single/Multiple Dose Escalation of TQC3721 Inhalation Powder in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Clinical Study of TQC3721 Inhalation Powder in Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQC3721-D8-I-01
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC3721 inhalation powder (Experimental): TQC3721 inhalation powder is administered as a single dose or continuously for 7 days.
  Interventions: Drug: TQC3721 inhalation powder
- Placebo for TQC3721 inhalation powder (Placebo Comparator): Placebo for TQC3721 inhalation powder inhalation is administered as a single dose or continuously for 7 days.
  Interventions: Drug: Placebo for TQC3721 inhalation powder

INTERVENTIONS:
Drug: TQC3721 inhalation powder — TQC3721 is a target inhibitor.
  Arms: TQC3721 inhalation powder
Drug: Placebo for TQC3721 inhalation powder — Placebo without drug substance.
  Arms: Placebo for TQC3721 inhalation powder

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose escalation, multicenter study design. The purpose is to evaluate the safety, tolerability, pharmacokinetics, and pharmacokinetic characteristics of TQC3721 inhalation powder in Chronic Obstructive Pulmonary Disease(COPD) patients with single/multiple dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-75 years old, male or female;
* During screening, according to the Global Oceanographic Library for Discovery (GOLD)guidelines (2024), patients diagnosed with stable moderate to severe COPD should have Force Expiratory Volume in 1 second (FEV1)/ forced vital capacity (FVC)<0.7 after inhaling bronchodilators; 40% ≤ FEV1 accounts for ≤ 80% of the expected value;
* When screening, after inhaling salbutamol aerosol for 4 times, there is a certain reversibility in the airway: the absolute value of FEV1 improves by more than 100ml;
* Being able to adjust the current COPD treatment or for COPD patients with initial treatment, prescribed bronchodilators, including Long-acting Muscarinic Antagonists (LAMA) and/or Long-acting β2-agonist (LABA) inhaled drugs, can be discontinued during the screening period after signing the informed consent form;
* The subject is able to discontinue Short acting Beta agonists (SABA) for at least 6 hours and Short acting Anticholinergic Agents (SAMA) for at least 8 hours;
* Smoking history ≥ 10 pack years (pack years: number of packs per day multiplied by smoking years);
* There is no evidence to suggest active respiratory and/or cardiovascular diseases other than COPD in clinical practice (such as uncontrolled hypertension);
* No other related lung diseases or history of thoracic surgery;
* The subjects were able to undergo reproducible FEV1 lung function testing according to the the American Thoracic Society and the European Respiratory Society (ATS/ERS) 2005 standard during screening;
* Body mass index (BMI) is between 18-30kg/m2;
* Participants must agree to use contraceptive methods (such as birth control pills, condoms, or intrauterine devices) with sexual partners of childbearing age during the clinical trial period (screening period to 30 days after the last dose);
* The subject is able to use a dry powder inhaler correctly for inhalation.
* Fully understand this study, voluntarily participate, and have signed the "Informed Consent Form".

Exclusion Criteria:

* History or current clinical instability of heart, respiratory, endocrine, metabolic, renal, liver, gastrointestinal, skin, infection, blood system, nervous system, or neurological/psychiatric disorders/abnormalities;
* The result of the human immunodeficiency virus (HIV) antibody test is positive; The result of hepatitis B surface antigen (HBsAg) test is positive (if HBsAg is positive, Hepatitis B virus deoxyribonucleic acid (HBV-DNA) should be checked if necessary, and if HBV-DNA<Lower Limit of Quantification (LLOQ), it does not need to be excluded); Hepatitis C virus (HCV) antibody positive and confirmed presence of HCV ribonucleic acid (RNA); Positive for Treponema pallidum antibody (TPPA);
* Have a history of illegal drug abuse in the past;
* Have participated in other clinical trials and received the investigational drug within 3 months prior to participating in this trial, or within 5 half lives of the investigational drug, whichever is shorter;
* Those who have lost blood or donated more than 400 mL of blood within 2 months before the experiment;
* Have any clear and severe history of drug or food allergies, especially those who are allergic to ingredients similar to the investigational drug;
* Drinking history (drinking 14 units of alcohol per week: 1 unit=285 ml of beer; or 25 ml of spirits; or 1 glass of wine);
* History of malignant tumors in any organ system within the past 5 years, regardless of whether treatment has been received or not, except for local basal cell carcinoma of the skin;
* Lower respiratory tract infection occurred within 6 weeks before screening or randomization. Upper respiratory tract infections requiring antibiotics within 6 weeks prior to screening or randomization;
* Have a history of active tuberculosis, bronchiectasis, asthma or other non-specific lung diseases.
* QT interval corrected using Fridericia's formula (QTcF)/R-wave peak to R-wave peak (RR [s]) interval, male>450ms, female>470ms, or history of long QT syndrome before screening or randomization;
* Subjects with a history of drug use in the past 2 years;
* Subjects who are unable to comply with past medication and concomitant medication restrictions;
* If there is a history of acute exacerbation of COPD within 3 months before screening or randomization, hospitalization or additional COPD maintenance treatment is required. Over the past three years, the average number of frequent exacerbations of COPD with moderate to severe severity has been ≥ 2 per year, or resulting in hospitalization for ≥ 2 acute exacerbations per year;
* Oral non selective beta blockers;
* Any situation that researchers believe may pose safety risks to subjects in the trial or may interfere with the conduct of this study, or where researchers believe that subjects may not be able to complete this study or may not be able to comply with the requirements of this study (due to management or other reasons).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | 19 days
  Incidence of adverse events (AE)
Serious Adverse Events (SAE) | 19 days
  Incidence of Serious Adverse Events (SAE)
Treatment-emergent adverse events (TEAEs) | 19 days
  Incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Plasma drug peak concentration | 9 days
  Plasma drug peak concentration after administration.
COPD Assessment Tes (CAT) scores | From day 1 to day 11 or end of treatment, whichever came first
  CAT score after administration. The score range is 0 to 40 points (0 to 10 is minor influence; 11 to 20 are moderate; 21 to 30 are classified as severe impact; 31 to 40 is very severe).

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China